CLINICAL TRIAL: NCT06387303
Title: Pain Control and Quality of Recovery After Intravenous Methadone Versus Intrathecal Morphine in Major Abdominal Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Priyanka Singla, Assistant Professor of Anesthesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSR230492
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Morphine

STUDY DESIGN:
Intervention Model Description: a single blind study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Morphine (Active Comparator): 250 mcg Intrathecal Injection prior to incision
  Interventions: Drug: Morphine
- Intravenous Methadone (Experimental): 0.2 mg / kg Intravenous delivery prior to incision. Maximum dosage will be 20 mg.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — Intravenous Methadone
  Other Names: Intrathecal Methadone
  Arms: Intravenous Methadone
Drug: Morphine — Intrathecal Morphine
  Other Names: Intravenous Morphine
  Arms: Intrathecal Morphine

SUMMARY:
Moderate to severe postoperative pain is relatively common after major abdominal surgery. It is associated with less than optimal surgical experience, poor quality of recovery, and the development of persistent postsurgical pain. Opioids remain a significant component of postoperative pain management. Side effects of opioids used for the treatment of postoperative pain include constipation, pruritus, nausea, and vomiting. Enhanced recovery after surgery (ERAS) protocols involve the utilization of multimodal analgesia. Analgesic techniques used include epidural analgesia, nerve blocks, and Intrathecal (IT) administration of morph ne. IT morphine reduces the postoperative opioid requirement for 18-24 hours after major abdominal surgery and reduces hospital length of stay (LOS) compared with epidural analgesia. A significant number of patients who receive IT morphine still experience moderate to severe postoperative p in. Additionally, many patients refuse the invasive procedure or cannot receive IT morphine due to procedure contraindications, thrombocytopenia, and/or coagulopathy.

Intravenous (IV) methadone has a long analgesic half-life and has N-methyl-D-aspartate (NMDA) receptor antagonist and serotonin and norepinephrine reuptake inhibitor (SNRI) properties. It has previously been shown to reduce postoperative opioid requirements, postoperative nausea and vomiting (PONV), and postoperative pain scores in patients who underwent orthopedic, abdominal, complex spine, and cardiac surg ry. Similar findings have been shown in obstetric patients who underwent cesarean delivery under general anesthesia as well as patients who underwent gynecologic surgery. IV methadone has, however, never been compared with IT morphine as a postoperative analgesic.

The hypothesis is that intravenous (IV) methadone is non-inferior to IT morphine in patients who undergo major abdominal surg ry. It offers the advantage of being a noninvasive analgesic modality that may contribute to decreasing opioid consumption during the first 72 hours postoperatively, controlling postoperative pain, and improving the quality of recovery after surgery.

DETAILED DESCRIPTION:
Moderate to severe postoperative pain is relatively common after major abdominal surgery. It is associated with less than optimal surgical experience, poor quality of recovery, and the development of persistent postsurgical pain. Opioids remain a significant component of postoperative pain management. Side effects of opioids used for the treatment of postoperative pain include constipation, pruritus, nausea, and vomiting. Enhanced recovery after surgery (ERAS) protocols involve the utilization of multimodal analgesia. Analgesic techniques used include epidural analgesia, nerve blocks, and Intrathecal (IT) administration of morph ne. IT morphine reduces the postoperative opioid requirement for 18-24 hours after major abdominal surgery and reduces hospital length of stay (LOS) compared with epidural analgesia. A significant number of patients who receive IT morphine still experience moderate to severe postoperative p in. Additionally, many patients refuse the invasive procedure or cannot receive IT morphine due to procedure contraindications, thrombocytopenia, and/or coagulopathy.

Intravenous (IV) methadone has a long analgesic half-life and has N-methyl-D-aspartate (NMDA) receptor antagonist and serotonin and norepinephrine reuptake inhibitor (SNRI) properties. It has previously been shown to reduce postoperative opioid requirements, postoperative nausea and vomiting (PONV), and postoperative pain scores in patients who underwent orthopedic, abdominal, complex spine, and cardiac surg ry. Similar findings have been shown in obstetric patients who underwent cesarean delivery under general anesthesia as well as patients who underwent gynecologic surgery. IV methadone has, however, never been compared with IT morphine as a postoperative analgesic.

The hypothesis is that intravenous (IV) methadone is non-inferior to IT morphine in patients who undergo major abdominal surg ry. It offers the advantage of being a noninvasive analgesic modality that may contribute to decreasing opioid consumption during the first 72 hours postoperatively, controlling postoperative pain, and improving the quality of recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an American Society of Anesthesiologists (ASA) physiological status I-III
* Undergoing laparotomy with midline incision
* Body mass index (BMI) between 18.5 and 45
* Ability to understand and read English
* Willingness and ability to comply with scheduled visits and study procedures

Exclusion Criteria:

* Not able or unwilling to sign consent
* Patients undergoing ambulatory surgery or anticipated to be discharged sooner than 24 hours after surgery
* Patients with chronic pain, requiring daily opioid use at the time of surgery, MME >60 as the FDA defines opioid tolerant as 60 MME, long-acting forms of opioids such as fentanyl patch, oxycontin.
* Pregnant Women
* Patients requiring emergent surgery
* Contraindications to neuraxial anesthesia including:

  * Coagulopathy
  * localized infection at the site of injection
  * pre-existing spinal pathology, specifically defined as active radiculopathy, severe central canal stenosis in the lumbar region, or an acute fracture in the lumbar region
* length of the QT interval (QTc) >450 on the most recent preoperative electrocardiogram (EKG)
* Prior spinal fusion
* Active or Prior Substance Use Disorder, undergoing active treatment with Medication of Opioid Use Disorder including methadone (once daily dosing), Buprenorphine (any formulation) and Naltrexone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 15 score | 24 hours, 48 hours, 72 hours, 42 days, 92 days
  The Quality of Recovery-15 (QoR-15) scale is a patient-reported outcome measurement of the quality of recovery after surgery and anesthesia. The scale ranges from 0 to 150, with a higher score indicating a better quality of recovery. A score of 0 indicates extremely poor quality of recovery, while a score of 150 indicates excellent quality of recovery. The QoR-15 score can be classified into four severity classes: excellent, good, moderate, and poor recovery.
Overall Benefits of Analgesic Score | 24 hours, 48 hours, 72 hours, 42 days, 92 days
  The overall benefit of analgesic score (OBAS) is a daily survey that assesses a patient's satisfaction with analgesia, pain intensity, and adverse effects.
  To compute score, add all scores in items 1-7. Range: [0 - 28]. A low score indicates high benefit
  1. Rate your current pain at rest on a scale between 0=minimal pain and 4=maximum imaginable pain
  2. Grade any distress and bother from vomiting in the past 24 hours (0=not at all to 4=very much)
  3. Grade any distress and bother from itching in the past 24 hours (0=not at all to 4=very much)
  4. Grade any distress and bother from sweating in the past 24 hours (0=not at all to 4=very much)
  5. Grade any distress and bother from freezing in the past 24 hours (0=not at all to 4=very much)
  6. Grade any distress and bother from dizziness in the past 24 hours (0=not at all to 4=very much)
  7. How satisfied are you with your pain treatment during the past 24 hours (0=not at all to 4= very much)
morphine milligram equivalent | 24 hours, 48 hours, 72 hours
  morphine milligram equivalent is a measurement of a given analgesic effect standardized to a milligram of morphine. In other words agent X has the same effect as Y milligrams of morphine.
Numeric Rating Scale pain scores (NRS) | 24 hours, 48 hours, 72 hours
  The numeric rating scale (NRS) is a pain screening tool commonly used to assess pain severity at a given moment in time. It uses a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."

SECONDARY OUTCOMES:
McGill Pain questionnaire score | 42 days, 92 days
  The McGill Pain Questionnaire (MPQ), also known as the McGill Pain Index, is a self-report questionnaire that helps patients describe the quality and intensity of their pain that assesses three components of pain experience: Sensory intensity, Emotional impact, and Cognitive evaluation of pain.
  The MPQ consists of 20 categories of verbal descriptors, 78 pain-related descriptors, and six words for current pain intensity. The descriptors fall into four major groups:
  Sensory: 1 to 10 Affective: 11 to 15 Evaluative: 16 Miscellaneous: 17 to 20 Each descriptor has a rank value based on its position in the word set. The sum of the rank values is the pain rating index (PRI). The maximum pain score is 78, and the higher the score, the greater the pain.
  The MPQ is valid, reliable, and sensitive for measuring cancer pain.
Numeric Rating Pain Score (NRS) | 42 days, 92 days
  The numeric rating scale (NRS) is a pain screening tool commonly used to assess pain severity at a given moment. It uses a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandsborg B, Nikolajsen L, Hansen CT, Kehlet H, Jensen TS. Risk factors for chronic pain after hysterectomy: a nationwide questionnaire and database study. Anesthesiology. 2007 May;106(5):1003-12. doi: 10.1097/01.anes.0000265161.39932.e8. PMID 17457133
- [Background] Bauchat JR, Habib AS. Evidence-based anesthesia for major gynecologic surgery. Anesthesiol Clin. 2015 Mar;33(1):173-207. doi: 10.1016/j.anclin.2014.11.011. Epub 2014 Dec 31. PMID 25701935
- [Background] Hein A, Rosblad P, Gillis-Haegerstrand C, Schedvins K, Jakobsson J, Dahlgren G. Low dose intrathecal morphine effects on post-hysterectomy pain: a randomized placebo-controlled study. Acta Anaesthesiol Scand. 2012 Jan;56(1):102-9. doi: 10.1111/j.1399-6576.2011.02574.x. PMID 22150410
- [Background] Modesitt SC, Sarosiek BM, Trowbridge ER, Redick DL, Shah PM, Thiele RH, Tiouririne M, Hedrick TL. Enhanced Recovery Implementation in Major Gynecologic Surgeries: Effect of Care Standardization. Obstet Gynecol. 2016 Sep;128(3):457-66. doi: 10.1097/AOG.0000000000001555. PMID 27500337
- [Background] Horlocker TT, Vandermeuelen E, Kopp SL, Gogarten W, Leffert LR, Benzon HT. Regional Anesthesia in the Patient Receiving Antithrombotic or Thrombolytic Therapy: American Society of Regional Anesthesia and Pain Medicine Evidence-Based Guidelines (Fourth Edition). Reg Anesth Pain Med. 2018 Apr;43(3):263-309. doi: 10.1097/AAP.0000000000000763. No abstract available. PMID 29561531
- [Background] Kharasch ED. Intraoperative methadone: rediscovery, reappraisal, and reinvigoration? Anesth Analg. 2011 Jan;112(1):13-6. doi: 10.1213/ANE.0b013e3181fec9a3. No abstract available. PMID 21173206
- [Background] Mancini I, Lossignol DA, Body JJ. Opioid switch to oral methadone in cancer pain. Curr Opin Oncol. 2000 Jul;12(4):308-13. doi: 10.1097/00001622-200007000-00006. PMID 10888415
- [Background] Slotkin TA, Seidler FJ, Whitmore WL. Methadone inhibits serotonin and norephinephrine uptake into rat brain synaptosomes and synaptic vesicles in vitro but not in vivo. Eur J Pharmacol. 1978 Jun 15;49(4):357-62. doi: 10.1016/0014-2999(78)90309-6. PMID 668807
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Machado FC, Palmeira CCA, Torres JNL, Vieira JE, Ashmawi HA. Intraoperative use of methadone improves control of postoperative pain in morbidly obese patients: a randomized controlled study. J Pain Res. 2018 Oct 2;11:2123-2129. doi: 10.2147/JPR.S172235. eCollection 2018. PMID 30323647
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Background] Russell T, Mitchell C, Paech MJ, Pavy T. Efficacy and safety of intraoperative intravenous methadone during general anaesthesia for caesarean delivery: a retrospective case-control study. Int J Obstet Anesth. 2013 Jan;22(1):47-51. doi: 10.1016/j.ijoa.2012.10.007. Epub 2012 Dec 7. PMID 23219678
- [Background] Richlin DM, Reuben SS. Postoperative pain control with methadone following lower abdominal surgery. J Clin Anesth. 1991 Mar-Apr;3(2):112-6. doi: 10.1016/0952-8180(91)90007-a. PMID 2039637
- [Background] Bergstrom JE, Scott ME, Alimi Y, Yen TT, Hobson D, Machado KK, Tanner EJ 3rd, Fader AN, Temkin SM, Wethington S, Levinson K, Sokolinsky S, Lau B, Stone RL. Narcotics reduction, quality and safety in gynecologic oncology surgery in the first year of enhanced recovery after surgery protocol implementation. Gynecol Oncol. 2018 Jun;149(3):554-559. doi: 10.1016/j.ygyno.2018.04.003. Epub 2018 Apr 13. PMID 29661495
- [Background] Krantz MJ, Martin J, Stimmel B, Mehta D, Haigney MC. QTc interval screening in methadone treatment. Ann Intern Med. 2009 Mar 17;150(6):387-95. doi: 10.7326/0003-4819-150-6-200903170-00103. Epub 2009 Jan 19. PMID 19153406